CLINICAL TRIAL: NCT00626431
Title: A Phase 3, Multi-Center, Open-Label, Trial to Evaluate the Efficacy, Safety and Pharmacokinetics of Two 6-Month Leuprolide Formulations, in Subjects With Prostatic Adenocarcinoma
Brief Title: A Study of Leuprolide to Treat Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Kristof Chwalisz, MD, PhD Therapeutic Area Head, Abbott
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: L-PC07-169
Record Dates: First submitted 2008-02-20; First posted 2008-02-29 (Estimated); Results first posted 2010-11-01 (Estimated); Last update posted 2011-07-19 (Estimated); Status verified 2011-07

CONDITIONS: Prostate Cancer
Keywords: Lupron Depot; prostate cancer; leuprolide acetate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Leuprolide acetate - Formulation A (Experimental): Leuprolide acetate 45 mg, 6-month depot
  Interventions: Drug: Leuprolide acetate - Formulation A
- Leuprolide acetate - Formulation B (Experimental): Leuprolide acetate, 45 mg, 6-month depot
  Interventions: Drug: Leuprolide acetate - Formulation B

INTERVENTIONS:
Drug: Leuprolide acetate - Formulation A — Leuprolide acetate was administered as 2 intramuscular (IM) injections of Formulation A, 45 mg 6 month depot, 24 weeks apart.
  Other Names: Lupron; leuprorelin; gonadotropin hormone-releasing hormone (GnRH); luteinizing hormone-releasing hormone (LHRH)
  Arms: Leuprolide acetate - Formulation A
Drug: Leuprolide acetate - Formulation B — Leuprolide acetate was administered as 2 intramuscular (IM) injections of Formulation B, 45 mg 6 month depot, 24 weeks apart.
  Other Names: Lupron; leuprorelin; gonadotropin hormone-releasing hormone (GnRH); luteinizing hormone-releasing hormone (LHRH)
  Arms: Leuprolide acetate - Formulation B

SUMMARY:
To assess the efficacy and safety of 2 new formulations of leuprolide acetate 45 mg 6-month depot, Formulation A or Formulation B, for the treatment of patients with prostate cancer. A formulation will be deemed successful if the percentage of subjects with suppression of testosterone to <= 50 ng/dL from Week 4 to Week 48 is not less than 87%, (the lower bound of the 2-sided 90% confidence interval), a protocol-specified criterion.

DETAILED DESCRIPTION:
A total of 300 male subjects were planned to be enrolled. Subjects were to receive a total of 2 intramuscular (IM) injections of the same formulation, either Formulation A or Formulation B, administered 24 weeks apart. The first 150 subjects were to receive Formulation A for both injections and the next 150 subjects were to receive Formulation B for both injections. The sponsor was to conduct an ongoing review of the primary endpoint data (suppression of testosterone <= 50 ng/dL) and planned to stop enrollment of Formulation A or Formulation B, or not to administer the second injection of Formulation A or Formulation B, if 15 or more subjects did not achieve testosterone suppression by Week 4 or failed to maintain testosterone suppression during the treatment period.

All analyses and summaries were to be conducted separately for subjects who received Formulation A or Formulation B.

This study was to be conducted at approximately 60-80 investigative sites. Subjects participated in the trial for approximately 14 months.

This trial was to include a Screening Period (up to 4 weeks), a 12-month Treatment Period (two 6-month treatment cycles), and a Follow-Up Period (30 days).

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily sign an IRB-approved informed consent form and any required privacy statement/authorization form.
* Pre-trial serum testosterone level >150 ng/dL.
* Histologically-confirmed prostatic adenocarcinoma in Jewett Clinical Stage A2, B, C or D and TNM* classification cT1b-4, N: any, M: any.

  *Tumor/Nodes/Metastases
* Subjects with a rising PSA following radical prostatectomy defined as an increase of 0.2 ng/mL from the previous test on two consecutive testings or rising PSA following prostate irradiation using Phoenix Definition of a rise of greater than or equal to 2.0 ng/mL above the nadir.
* Prostate cancer and general clinical status is sufficient to warrant at least 48 weeks of continuous androgen deprivation treatment, without concomitant antiandrogen treatment.
* Eastern Cooperative Oncology Group (ECOG) Performance status grades 0,1,or 2 at the time of pre-trial screening.
* Life expectancy of at least 18 months.
* Subjects with serum creatinine ≤1.9 mg/dL, bilirubin ≤2.0 mg/dL (unless Gilbert's syndrome with normal AST, ALT); AST and ALT ≤2.5 times the upper limit of normal.

Exclusion Criteria:

* Requires additional treatment including radical prostatectomy, radiotherapy or cryotherapy of local disease.
* Historical, clinical, or radiographic evidence of central nervous system metastases, including spinal cord metastasis.
* Clinical evidence of urinary tract obstruction.
* History of bilateral orchiectomy, adrenalectomy, or hypophysectomy.
* History of clinical hypogonadism.
* Current malignancy or history of malignancy except for prostate cancer or basal or squamous cell carcinoma of the skin.
* Clinical or laboratory evidence of any severe underlying disease state (excluding prostate cancer) that would place subjects in additional jeopardy by participating in this trial.
* Hypersensitivity to leuprolide, polylactic acid, or any excipient of the drug.
* Incomplete recovery from the effects of any major surgery.
* History of receiving of the following prostate cancer therapies within 8 weeks prior to the Screening Visit: chemotherapy, immunotherapy, antiandrogen, radiation therapy, cryotherapy, strontium, or biological response modifiers.
* History of prostatic surgery within 4 weeks prior to the Screening Visit.
* Received hormonal therapy, including GnRH analogs (less than or equal to 6 month depot administration), estrogen, Megace and phytotherapy, within 32 weeks prior to the Screening Visit and during the trial.
* Alternative medical therapies which have an estrogenic, androgenic, or antiandrogenic effect (including phyto-estrogens and phyto-androgens) within 12 weeks prior to the Screening Visit and during the trial.
* Requires the chronic use of systemic corticosteroids and anticonvulsants that may affect bone loss such as carbamazepine, phenobarbital, phenytoin, valproic acid or primidone.
* May require antiandrogen, immuno-, or surgical therapy for prostate cancer during the trial.
* History of alcoholism or consumes >14 alcoholic beverages per week or illicit drug abuse within 12 months prior to screening.
* Received therapy with a GnRH analog (1 year implant) within 60 weeks prior to the Screening Visit.
* Received therapy with finasteride or ketoconazole within 1 week prior to the Screening Visit; dutasteride within 25 weeks prior to the Screening Visit.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2008-02; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristof Chwalisz, MD, PhD, Study Director — Abbott
Locations (63):
- United States (63):
  - Site Reference ID/Investigator# 8696, Birmingham, Alabama
  - Site Reference ID/Investigator# 8681, Homewood, Alabama
  - Site Reference ID/Investigator# 8569, Anchorage, Alaska
  - Site Reference ID/Investigator# 9709, Phoenix, Arizona
  - Site Reference ID/Investigator# 8662, Sierra Vista, Arizona
  - Site Reference ID/Investigator# 8656, Tucson, Arizona
  - Site Reference ID/Investigator# 9705, Little Rock, Arkansas
  - Site Reference ID/Investigator# 8691, Anaheim, California
  - Site Reference ID/Investigator# 8566, Atherton, California
  - Site Reference ID/Investigator# 8686, Fresno, California
  - Site Reference ID/Investigator# 8698, Laguna Hills, California
  - Site Reference ID/Investigator# 9703, Long Beach, California
  - Site Reference ID/Investigator# 8674, Los Angeles, California
  - Site Reference ID/Investigator# 8650, Tarzana, California
  - Site Reference ID/Investigator# 8699, Torrance, California
  - Site Reference ID/Investigator# 8668, Denver, Colorado
  - Site Reference ID/Investigator# 8646, Englewood, Colorado
  - Site Reference ID/Investigator# 8652, Middlebury, Connecticut
  - Site Reference ID/Investigator# 8697, New Britain, Connecticut
  - Site Reference ID/Investigator# 8655, Aventura, Florida
  - Site Reference ID/Investigator# 8648, Daytona Beach, Florida
  - Site Reference ID/Investigator# 8660, New Smyrna Beach, Florida
  - Site Reference ID/Investigator# 8658, Orange City, Florida
  - Site Reference ID/Investigator# 8664, Orlando, Florida
  - Site Reference ID/Investigator# 8651, Saint Augustine, Florida
  - Site Reference ID/Investigator# 8661, St. Petersburg, Florida
  - Site Reference ID/Investigator# 8568, Tallahassee, Florida
  - Site Reference ID/Investigator# 8679, Wellington, Florida
  - Site Reference ID/Investigator# 8562, West Palm Beach, Florida
  - Site Reference ID/Investigator# 8670, Roswell, Georgia
  - Site Reference ID/Investigator# 9708, Thomasville, Georgia
  - Site Reference ID/Investigator# 8693, Fort Wayne, Indiana
  - Site Reference ID/Investigator# 8690, Newburgh, Indiana
  - Site Reference ID/Investigator# 8565, Overland Park, Kansas
  - Site Reference ID/Investigator# 8676, Greenbelt, Maryland
  - Site Reference ID/Investigator# 8653, Las Vegas, Nevada
  - Site Reference ID/Investigator# 8667, Lawrenceville, New Jersey
  - Site Reference ID/Investigator# 8665, New York, New York
  - Site Reference ID/Investigator# 8657, Poughkeepsie, New York
  - Site Reference ID/Investigator# 9702, The Bronx, New York
  - Site Reference ID/Investigator# 8680, Charlotte, North Carolina
  - Site Reference ID/Investigator# 8673, Concord, North Carolina
  - Site Reference ID/Investigator# 8666, Raleigh, North Carolina
  - Site Reference ID/Investigator# 8570, Salisbury, North Carolina
  - Site Reference ID/Investigator# 8644, Winston-Salem, North Carolina
  - Site Reference ID/Investigator# 8663, Cincinnati, Ohio
  - Site Reference ID/Investigator# 8567, Columbus, Ohio
  - Site Reference ID/Investigator# 8678, Bethany, Oklahoma
  - Site Reference ID/Investigator# 8563, Bala-Cynwyd, Pennsylvania
  - Site Reference ID/Investigator# 8692, Lancaster, Pennsylvania
  - Site Reference ID/Investigator# 8689, Myrtle Beach, South Carolina
  - Site Reference ID/Investigator# 8643, Germantown, Tennessee
  - Site Reference ID/Investigator# 8695, Germantown, Tennessee
  - Site Reference ID/Investigator# 8685, Memphis, Tennessee
  - Site Reference ID/Investigator# 8564, Nashville, Tennessee
  - Site Reference ID/Investigator# 8645, Nashville, Tennessee
  - Site Reference ID/Investigator# 8641, Dallas, Texas
  - Site Reference ID/Investigator# 8675, Houston, Texas
  - Site Reference ID/Investigator# 8684, San Antonio, Texas
  - Site Reference ID/Investigator# 8649, Tyler, Texas
  - Site Reference ID/Investigator# 8683, Salt Lake City, Utah
  - Site Reference ID/Investigator# 8672, Norfolk, Virginia
  - Site Reference ID/Investigator# 8669, Richmond, Virginia

REFERENCES:
- [Derived] Spitz A, Young JM, Larsen L, Mattia-Goldberg C, Donnelly J, Chwalisz K. Efficacy and safety of leuprolide acetate 6-month depot for suppression of testosterone in patients with prostate cancer. Prostate Cancer Prostatic Dis. 2012 Mar;15(1):93-9. doi: 10.1038/pcan.2011.50. Epub 2011 Oct 25. PMID 22025196

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The enrollment of subjects with Formulation A occurred sequentially before the enrollment of subjects with Formulation B.
Pre-assignment Details: Formulation A and Formulation B treatment groups were enrolled sequentially. All analyses and summaries were conducted separately for both treatment groups.
Groups:
- Leuprolide Acetate - Formulation A: Leuprolide acetate 45 mg, 6-month depot administered as 2 intramuscular (IM) injections of Formulation A, 24 weeks apart. Injections were administered on Day 1 and Day 169. The first 150 subjects were to receive Formulation A and then the next 150 subjects were to receive Formulation B in a sequential manner.
- Leuprolide Acetate - Formulation B: Leuprolide acetate 45 mg, 6-month depot administered as 2 intramuscular injections of Formulation B, 24 weeks apart. Injections were administered on Day 1 and Day 169. The first 150 subjects were to receive Formulation A and then the next 150 subjects were to receive Formulation B in a sequential manner.
Period: Overall Study
Arm/Group | Leuprolide Acetate - Formulation A | Leuprolide Acetate - Formulation B
Started | 151 (Separate groups of subjects received Formulation A and B and data were not compared between groups.) | 159 (Separate groups of subjects received Formulation A and B and data were not compared between groups.)
Completed | 134 | 114
Not Completed | 17 | 45

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leuprolide Acetate - Formulation A | Leuprolide Acetate - Formulation B | Total
Number analyzed (Participants) | 151 | 159 | 310
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 33 | 51
  >=65 years | 133 | 126 | 259
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 151 | 159 | 310
Region of Enrollment [Number; unit: participants]
  United States | 151 | 159 | 310

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Suppression of Serum Testosterone (<=50 ng/dL) From Week 4 to Week 48 for Formulation A: Intent-to-treat (ITT) Population for the Primary Endpoint.
Description: The percentage of subjects with testosterone suppression (<= 50 ng/dL) from Week 4 to Week 48 was calculated by the Kaplan-Meier method for right-censored observations. Subjects who failed testosterone suppression were considered failures on the first day of a testosterone measurement (>50 ng/dL). Subjects who prematurely discontinued without escaping and those who were successfully suppressed through Week 48 were censored at their last measured testosterone value (Day 337 to Day 340 at Week 48). The 90% 2-sided confidence interval was calculated from Kaplan-Meier estimates.
Time Frame: Week 4 to Week 48
Population: The ITT population for the primary endpoint was the same as the ITT population for the secondary endpoints and also excluded subjects whose final testosterone values were measured before Day 19 without suppression (>50 ng/dL) or whose testosterone levels remained suppressed through Week 48 but testosterone levels were not measured at Week 4.
Measure: Number (90% Confidence Interval); unit: Percent Suppressed
Groups:
- Leuprolide Acetate - Formulation A: Leuprolide acetate 45 mg, 6-month depot administered as 2 intramuscular injections of Formulation A, 24 weeks apart. Injections were administered on Day 1 and Day 169. The first 150 subjects were to receive Formulation A and then the next 150 subjects were to receive Formulation B in a sequential manner.
Arm/Group | Leuprolide Acetate - Formulation A
Number analyzed (Participants) | 148
Percent Suppressed | 93.6 (2.05) [90.2 to 97.0]

2. Secondary Outcome: Mean Testosterone Concentration (+/- Standard Error) at Each Visit for Formulation A: ITT Population
Description: Baseline was the last measurement before the first dose of Formulation A. The mean +/- standard error was calculated at each visit. The final visit occurred at Week 48 unless the subject prematurely discontinued the study.
Time Frame: Baseline, Days 2 and 8, Weeks 2, 4, 8, 14, 20, 24, 26, 30, 34, 40, 46, 48, and Final Visit
Population: The ITT population included subjects who received at least 1 dose of study drug, who had at least 1 postbaseline measurement, and who did not use prohibited medications during the first 32 days after the initiation of study drug treatment that either lowered testosterone levels or blocked its action.
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Leuprolide Acetate - Formulation A
Number analyzed (Participants) | 151
ng/dL
  Testosterone concentration at baseline | 432.9 (14.35)
  Testosterone concentration at Day 2 | 613.1 (21.53)
  Testosterone concentration at Day 8 | 468.2 (16.55)
  Testosterone concentration at Week 2 | 127.1 (7.36)
  Testosterone concentration at Week 4 | 16.0 (0.70)
  Testosterone concentration at Week 8 | 9.6 (0.46)
  Testosterone concentration at Week 14 | 9.2 (0.46)
  Testosterone concentration at Week 20 | 8.5 (0.46)
  Testosterone concentration at Week 24 | 14.3 (1.25)
  Testosterone concentration at Week 26 | 9.0 (0.47)
  Testosterone concentration at Week 30 | 9.9 (1.67)
  Testosterone concentration at Week 34 | 13.0 (4.14)
  Testosterone concentration at Week 40 | 8.8 (0.41)
  Testosterone concentration at Week 46 | 8.8 (0.46)
  Testosterone concentration at Week 48/Final Visit | 13.3 (3.67)

3. Secondary Outcome: Mean Testosterone Concentration (+/- Standard Error) at Each Visit for Formulation B: ITT Population
Description: Baseline was the last measurement before the first dose of Formulation B. The mean +/- standard error was calculated at each visit. The final visit occurred at Week 48 unless the subject prematurely discontinued the study.
Time Frame: Baseline, Days 2 and 8, Weeks 2, 4, 8, 14, 20, 24, 26, 30, 34, 40, 46, 48, and Final Visit
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Leuprolide Acetate - Formulation B
Number analyzed (Participants) | 157
ng/dL
  Testosterone concentration at baseline | 414.0 (14.15)
  Testosterone concentration at Day 2 | 578.0 (20.14)
  Testosterone concentration at Day 8 | 466.9 (17.70)
  Testosterone concentration at Week 2 | 127.4 (7.35)
  Testosterone concentration at Week 4 | 15.3 (0.71)
  Testosterone concentration at Week 8 | 9.1 (0.44)
  Testosterone concentration at Week 14 | 8.9 (0.42)
  Testosterone concentration at Week 20 | 9.6 (0.54)
  Testosterone concentration at Week 24 | 28.0 (3.97)
  Testosterone concentration at Week 26 | 15.6 (2.63)
  Testosterone concentration at Week 30 | 9.4 (0.60)
  Testosterone concentration at Week 34 | 9.7 (0.53)
  Testosterone concentration at Week 40 | 9.5 (0.52)
  Testosterone concentration at Week 46 | 9.4 (0.64)
  Testosterone concentration at Week 48/Final Visit | 13.8 (1.87)

4. Secondary Outcome: Mean (+/- Standard Error) Acute-on-chronic Changes in Testosterone From Pre-injection Levels for Formulation A: ITT Population
Description: The acute-on-chronic effect is an agonistic stimulation of serum testosterone after the second depot injection of Formulation A. The mean +/- standard error changes were measured to assess this effect from just before to 2 weeks after the second injection.
Time Frame: Week 24 before the second injection until 2 weeks after Week 24 (2 hours [h], 4 h, 8 h, 1 day [d], 2 d, 3-10 d, and 11-17 d postdose)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Leuprolide Acetate - Formulation A
Number analyzed (Participants) | 135
ng/dL
  Testosterone concentration at 2 hours postdose | -1.9 (0.85)
  Testosterone concentration at 4 hours postdose | -1.2 (0.93)
  Testosterone concentration at 8 hours postdose | -1.3 (1.02)
  Testosterone concentration at Day 1 postdose | -0.1 (0.95)
  Testosterone concentration at Day 2 postdose | -0.1 (0.92)
  Testosterone concentration at Days 3-10 postdose | -1.0 (0.89)
  Testosterone concentration at Days 11-17 postdose | -2.1 (0.87)

5. Secondary Outcome: Mean (+/- Standard Error) Acute-on-chronic Changes in Testosterone From Pre-injection Levels for Formulation B: ITT Population
Description: The acute-on-chronic effect is an agonistic stimulation of serum testosterone after the second depot injection of Formulation B. The mean +/- standard error changes were measured to assess this effect from just before to 2 weeks after the second injection.
Time Frame: Week 24 before the second injection until 2 weeks after Week 24 (2 h, 4 h, 8 h, 1 d, 2 d, 3-10 d, and 11-17 d postdose)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Leuprolide Acetate - Formulation B
Number analyzed (Participants) | 124
ng/dL
  Testosterone concentration at 2 hours postdose | -0.7 (0.66) [-101.2 to 18.0]
  Testosterone concentration at 4 hours postdose | 1.6 (1.13) [-99.3 to 34.0]
  Testosterone concentration at 8 hours postdose | 3.6 (1.35) [-101.5 to 47.0]
  Testosterone concentration at Day 1 postdose | 8.0 (1.80) [-99.8 to 46.0]
  Testosterone concentration at Day 2 postdose | 7.8 (1.81) [-99.2 to 48.7]
  Testosterone concentration at Days 3-10 postdose | 4.5 (1.07) [-96.7 to 44.7]
  Testosterone concentration at Day 11-17 postdose | -4.2 (1.43) [-97.5 to 13.0]

6. Primary Outcome: Adjusted Percentage of Subjects With Suppression of Serum Testosterone (<=50 ng/dL) From Week 4 to Week 48 for Formulation A: ITT Population for the Primary Endpoint Adjusted
Description: The adjusted percentage of subjects with testosterone suppression (<= 50 ng/dL) from Week 4 to Week 48 was calculated by the Kaplan-Meier method for right-censored observations. The primary efficacy analysis was adjusted to censor subjects who received an anti-androgen at the last testosterone measurement before use of the anti-androgen. One additional subject was censored because of a laboratory error, at the last measurement before the error. The adjusted 90% 2-sided confidence interval was calculated from Kaplan-Meier estimates.
Time Frame: Week 4 to Week 48
Measure: Number (90% Confidence Interval); unit: Percent Suppressed
Arm/Group | Leuprolide Acetate - Formulation A
Number analyzed (Participants) | 148
Percent Suppressed | 93.4 [89.9 to 96.9]

7. Secondary Outcome: Mean (+/- Standard Error) Acute-on-chronic Changes in Luteinizing Hormone From Pre-injection Levels for Formulation A: ITT Population
Description: The acute-on-chronic effect is an agonistic stimulation of luteinizing hormone after the second depot injection of Formulation A. The mean +/- standard error changes were measured to assess this effect from just before to 2 weeks after the second injection.
Time Frame: Week 24 before the second injection until 2 weeks after Week 24 (2 h, 4 h, 8 h, 1 d, 2 d, 3-10 d, and 11-17 d postdose)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Leuprolide Acetate - Formulation A
Number analyzed (Participants) | 134
ng/dL
  Testosterone concentration at 2 hours postdose | 0.2 (0.03)
  Testosterone concentration at 4 hours postdose | 0.2 (0.03)
  Testosterone concentration at 8 hours postdose | 0.2 (0.02)
  Testosterone concentration at Day 1 postdose | 0.2 (0.02)
  Testosterone concentration at Day 2 postdose | 0.1 (0.01)
  Testosterone concentration at Days 3-10 postdose | 0.1 (0.01)
  Testosterone concentration at Days 11-17 postdose | 0.1 (0.02)

8. Secondary Outcome: Mean (+/- Standard Error) Acute-on-chronic Changes in Luteinizing Hormone From Pre-injection Levels for Formulation B: ITT Population
Description: The acute-on-chronic effect is an agonistic stimulation of luteinizing hormone after the second depot injection of Formulation B. The mean +/- standard error changes were measured to assess this effect from just before to 2 weeks after the second injection.
Time Frame: Week 24 before the second injection until 2 weeks after Week 24 (2 h, 4 h, 8 h, 1 d, 2 d, 3-10 d, and 11-17 d postdose)
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/dL
Arm/Group | Leuprolide Acetate - Formulation B
Number analyzed (Participants) | 123
ng/dL
  Testosterone concentration at 2 hours postdose | 0.4 (0.07)
  Testosterone concentration at 4 hours postdose | 0.5 (0.12)
  Testosterone concentration at 8 hours postdose | 0.4 (0.11)
  Testosterone concentration at Day 1 postdose | 0.4 (0.08)
  Testosterone concentration at Day 2 postdose | 0.2 (0.04)
  Testosterone concentration at Days 3-10 postdose | 0.1 (0.02)
  Testosterone concentration at Days 11-17 postdose | -0.1 (0.04)

9. Secondary Outcome: Mean (+/- Standard Error) Prostate Specific Antigen (PSA) at Baseline, Visits Throughout the Study, and at Final Visit for Formulation A: ITT Population
Description: PSA levels were measured at baseline and each treatment visit for Formulation A. The mean (+/- standard error) was calculated at each visit. The final visit occurred at Week 48 unless the subject prematurely discontinued the study.
Time Frame: Baseline, Day 8, Week 14, Week 24, Week 30, Week 40, Week 48, and the Final Visit
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Leuprolide Acetate - Formulation A
Number analyzed (Participants) | 151
ng/mL
  PSA concentration at baseline | 35.0 (11.21)
  PSA Concentration at Day 8 | 40.4 (12.90)
  PSA Concentration at Week 14 | 2.4 (0.62)
  PSA Concentration at Week 24 | 2.9 (1.09)
  PSA Concentration at Week 30 | 1.6 (0.46)
  PSA Concentration at Week 40 | 2.2 (0.82)
  PSA Concentration at Week 48/Final Visit | 3.7 (1.51)

10. Secondary Outcome: Mean (+/- Standard Error) Prostate Specific Antigen (PSA) at Baseline, Visits Throughout the Study, and at Final Visit for Formulation B: ITT Population
Description: PSA levels were measured at baseline and each treatment visit for Formulation B. The mean (+/- standard error) was calculated at each visit. The final visit occurred at Week 48 unless the subject prematurely discontinued the study.
Time Frame: Baseline, Day 8, Week 14, Week 24, Week 30, Week 40, Week 48, and the Final Visit
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Leuprolide Acetate - Formulation B
Number analyzed (Participants) | 157
ng/mL
  PSA concentration at baseline | 20.5 (3.88)
  PSA Concentration at Day 8 | 23.1 (4.03)
  PSA Concentration at Week 14 | 2.4 (0.51)
  PSA Concentration at Week 24 | 2.5 (0.65)
  PSA Concentration at Week 30 | 2.7 (0.86)
  PSA Concentration at Week 40 | 2.5 (0.85)
  PSA Concentration at Week 48/Final Visit | 6.2 (2.75)

11. Primary Outcome: Percentage of Subjects With Suppression of Serum Testosterone (<=50 ng/dL) From Week 4 to Week 48 for Formulation B: ITT Population for the Primary Endpoint Preplanned
Description: as for outcome 1
Time Frame: Week 4 to Week 48
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: Percent suppressed
Arm/Group | Leuprolide Acetate - Formulation B
Number analyzed (Participants) | 154
Percent suppressed | 86.9 [82.2 to 91.7]

ADVERSE EVENTS:
Time Frame: Both serious adverse events and adverse events were reported from the receipt of the first dose of study drug through the 30-day follow-up period.
Description: This study included 2 treatment groups, Formulation A or Formulation B. Summaries were conducted separately for both treatment groups and no statistical tests were performed between treatment groups.
Arm/Group | Leuprolide Acetate - Formulation A | Leuprolide Acetate - Formulation B
Serious Adverse Events (participants affected / at risk) | 31/151 | 41/159
Other Adverse Events (participants affected / at risk) | 133/151 | 127/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate - Formulation A (N=151) | Leuprolide Acetate - Formulation B (N=159)
anemia (Blood and lymphatic system disorders) | 2 | 0
acute coronary syndrome (Cardiac disorders) | 1 | 0
angina pectoris (Cardiac disorders) | 1 | 0
angina unstable (Cardiac disorders) | 1 | 1
atrial fibrillation (Cardiac disorders) | 2 | 0
atrioventricular block complete (Cardiac disorders) | 1 | 0
atrioventricular block second degree (Cardiac disorders) | 1 | 0
cardiac failure congestive (Cardiac disorders) | 2 | 3
coronary artery disease (Cardiac disorders) | 3 | 2
sick sinus syndrome (Cardiac disorders) | 1 | 0
iron deficiency anemia (Blood and lymphatic system disorders) | 0 | 1
acute myocardial infarction (Cardiac disorders) | 0 | 1
myocardial infarction (Cardiac disorders) | 0 | 1
palpitations (Cardiac disorders) | 0 | 1
ventricular tachycardia (Cardiac disorders) | 0 | 1
colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
fecaloma (Gastrointestinal disorders) | 0 | 1
intestinal perforation (Gastrointestinal disorders) | 0 | 1
esophageal achalasia (Gastrointestinal disorders) | 0 | 1
pancreatitis (Gastrointestinal disorders) | 0 | 1
pancreatitis acute (Gastrointestinal disorders) | 0 | 1
pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
retroperitoneal hemorrhage (Gastrointestinal disorders) | 1 | 0
vomiting (Gastrointestinal disorders) | 1 | 0
asthenia (General disorders) | 1 | 0
chest pain (General disorders) | 1 | 0
multi-organ failure (General disorders) | 0 | 1
cholecystitis (Hepatobiliary disorders) | 0 | 1
acute sinusitis (Infections and infestations) | 0 | 1
bronchiectasis (Infections and infestations) | 1 | 0
bronchitis (Infections and infestations) | 0 | 1
cellulitis (Infections and infestations) | 1 | 0
enterobacter sepsis (Infections and infestations) | 1 | 0
gastroenteritis (Infections and infestations) | 0 | 1
lobar pneumonia (Infections and infestations) | 1 | 1
pneumonia (Infections and infestations) | 2 | 3
septic shock (Infections and infestations) | 0 | 1
urinary tract infection (Infections and infestations) | 1 | 1
urosepsis (Infections and infestations) | 0 | 1
humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
in-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
rib fracture (Injury, poisoning and procedural complications) | 1 | 0
lung injury (Injury, poisoning and procedural complications) | 0 | 1
wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
hypoglycemia (Metabolism and nutrition disorders) | 1 | 0
hypovolemia (Metabolism and nutrition disorders) | 1 | 0
diabetic ketacidosis (Metabolism and nutrition disorders) | 0 | 1
arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
B-cell small lymphocytic lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
bladder cancer stage I, without cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
colon cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
non-Hodgkin's lymphoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
carotid artery stenosis (Nervous system disorders) | 2 | 0
cerebrovascular accident (Nervous system disorders) | 1 | 2
cerebrovascular disorder (Nervous system disorders) | 0 | 1
dementia (Nervous system disorders) | 0 | 1
hemorrhagic transformation stroke (Nervous system disorders) | 0 | 1
presyncope (Nervous system disorders) | 0 | 1
spinal hematoma (Nervous system disorders) | 1 | 0
syncope (Nervous system disorders) | 0 | 3
transient ischemic attack (Nervous system disorders) | 2 | 0
completed suicide (Psychiatric disorders) | 0 | 1
mental status change (Nervous system disorders) | 0 | 1
hematuria (Renal and urinary disorders) | 1 | 0
renal failure acute (Renal and urinary disorders) | 1 | 1
ureteric obstruction (Renal and urinary disorders) | 0 | 1
urinary retention (Renal and urinary disorders) | 0 | 1
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
hemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pleural effusion (Renal and urinary disorders) | 0 | 2
pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2
aortic aneurysm (Vascular disorders) | 1 | 0
deep vein thrombosis (Vascular disorders) | 0 | 1
hypotension (Vascular disorders) | 0 | 1
orthostatic hypotension (Vascular disorders) | 1 | 0
cholelithiasis (Hepatobiliary disorders) | 2 | 0
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprolide Acetate - Formulation A (N=151) | Leuprolide Acetate - Formulation B (N=159)
Anemia (Blood and lymphatic system disorders) | 6 | 9
constipation (Gastrointestinal disorders) | 15 | 16
nausea (Gastrointestinal disorders) | 5 | 8
fatigue (General disorders) | 18 | 14
injection site pain (General disorders) | 27 | 26
edema peripheral (General disorders) | 7 | 9
nasopharyngitis (Infections and infestations) | 10 | 15
upper respiratory tract infection (Infections and infestations) | 8 | 9
urinary tract infection (Infections and infestations) | 7 | 8
arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 22
back pain (Musculoskeletal and connective tissue disorders) | 8 | 9
pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 9
insomnia (Psychiatric disorders) | 13 | 9
dizziness (Nervous system disorders) | 8 | 15
headache (Nervous system disorders) | 11 | 9
dysuria (Renal and urinary disorders) | 9 | 8
hematuria (Renal and urinary disorders) | 9 | 1
nocturia (Renal and urinary disorders) | 8 | 4
cough (Respiratory, thoracic and mediastinal disorders) | 10 | 6
dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 8
hot flush (Vascular disorders) | 88 | 71
hypertension (Vascular disorders) | 9 | 15
musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 8 | 6
rash (Skin and subcutaneous tissue disorders) | 9 | 6

LIMITATIONS AND CAVEATS:
Treatment with Formulation B was prematurely discontinued as testosterone was not adequately suppressed to <= 50 ng/dL or escapes from suppression occurred. Subjects who had not received dose 2 of Formulation B were discontinued after Week 24.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication, whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.